CLINICAL TRIAL: NCT01046448
Title: The Cardiovascular Morbidity in Children With Chronic Renal Failure Study
Brief Title: The Cardiovascular Comorbidity in Children With Chronic Kidney Disease Study
Acronym: 4C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: KfH Foundation for Preventive Medicine (Unknown); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Prof. Dr. med. Dr. h.c. Franz Schaefer, Center for Paediatrics and Adolescent Medicine, University of Heidelberg, Heidelberg, Germany
Other Study IDs: S-32/2009
Record Dates: First submitted 2009-08-07; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Kidney Disease; Pediatric; Cardiovascular Disease
Keywords: Children; chronic renal failure; chronic kidney disease; cardiovascular disease; cardiovascular morbidity; left ventricular hypertrophy; carotid intima media thickness; arterial stiffness; pulse wave velocity; augmentation index; left ventricular cardiac function; progression; genetic risk factors; vasculopathy; cardiopathy; whole genome analysis; haplotype analysis; SNP-screening
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Kidney Failure, Chronic; Hypertrophy, Left Ventricular; Disease Progression; Vascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, whole blood, urine, DNA, vessel biopsies,
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 4C: Children with chronic kidney disease stage IIIb to V (GFR 10 to 45 ml/min/1.73m²) at screening.

SUMMARY:
Children and adolescents with chronic kidney disease (CKD) are at high risk for cardiovascular (CV) morbidity and mortality. Recent studies suggest that pediatric patients with even moderately impaired kidney function may be afflicted with significant early cardiac and vascular abnormalities.

The pathogenesis and the natural course of CV comorbidity in pediatric CKD patients is still elusive. In this multicenter, prospective, observational study the prevalence, degree and progression of CV comorbidity in children will be characterized and related to CKD progression. The morphology and function of the heart and vessels will be monitored by sensitive, non-invasive methods and will be compared with aged matched healthy controls. Multiple potential clinical, anthropometric, biochemical, and pharmacological risk factors will be monitored prospectively and will be related to CV status. Genotyping might identify predisposing genetic factors for progression of CV comorbidity and underlying nephropathies.

DETAILED DESCRIPTION:
Adult patients with CKD are at markedly increased risk of dying from cardiovascular events. The risk is most dramatically increased in young patients with end-stage renal disease, who are almost as likely to die from cardiovascular causes as elderly individuals in the general population.

Early morphological and functional vascular abnormalities can be detected even in adolescents with CKD, but information about the prevalence, severity and natural course of vascular lesions in different stages of renal failure is lacking and the factors predisposing to an early onset and rapid progression of cardiovascular morbidity are still elusive.

The pediatric population appears uniquely suited to study the effects of CKD on the cardiovascular system due to the virtual absence of vascular morbidity related to ageing, diabetes and smoking.

In order to improve our understanding of the causes and consequences of cardiovascular comorbidity in children with progressive CKD, a consortium of pediatric nephrologists in Europe has joined to perform a long-term prospective observational study following the cardiovascular health of children as they advance through successive stages of CKD.

The 4C Study will follow up at least 625 patients aged 6 to 17 years with a glomerular filtration rate of 10 to 45 ml/min/1.73 m² in more than 40 pediatric nephrology units in 14 European countries.

The morphology and function of the heart and the large arteries is regularly assessed by sensitive, non-invasive methods and the findings compared to a large group of healthy children.

Multiple potential clinical, anthropometric, biochemical, and pharmacological risk factors are monitored prospectively and will be related to the cardiovascular status of the patients.

A whole genome association study will be performed to identify genetic variants associated with the progression of cardio-vascular alterations and renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 17 years
* GFR 10 to 45 ml/min/1.73m² (CKD stage IIIb to V);

Exclusion Criteria:

* Active systemic vasculitis
* Diabetes mellitus
* Renal vascular anomalies
* Anomalies of the limbs preventing standardized diagnostic procedures

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 650 children with CKD stage IIIb to V (GFR 10-45 ml/min/1.73m²). Children who reach end-stage renal disease will be continuously followed while on renal replacement therapy.
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Functional and morphological evidence of cardiovascular disease progression (arterial stiffness, myocardial dysfunction, cIMT, LVMI) and association with clinical, anamnestic, anthropometric, biochemical, drug-related and genetic risk factors | 3 years

SECONDARY OUTCOMES:
Genetic risk factors for early manifesting progressive vascular lesions and progressive kidney disease by the genome-wide SNP-screening and haplotype analysis. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Franz Schaefer, MD, Principal Investigator — Center for Pediatric and Adolescent Medicine, University of Heidelberg, Germany; Uwe Querfeld, MD, Principal Investigator — Klinik für Pädiatrie m.S. Nephrologie, Charite, 13353 Berlin, Germany
Locations (50):
- Medical University of Vienna, Vienna, Austria
- UZ Gent, Ghent, Belgium
- University Hospital Motol, Prague, Czechia
- France (2):
  - Service de Pédiatrie & Inserm U820, Lyon
  - Hôpital de Hautepierre, Strasbourg
- Germany (12):
  - Charité Children's Hospital, Berlin
  - University Children's Hospital, Cologne
  - University Children's Hospital, Erlangen
  - University Children's Hospital, Essen
  - Center for Pediatrics and Adolescent Medicine, Freiburg im Breisgau
  - UKE University Children's Hospital, Hamburg
  - Hannover Medical School, Hanover
  - Center for Pediatrics and Adolescent Medicine, Heidelberg
  - City Hospital St. Georg, Leipzig
  - KfH Kidney Center for Children, Marburg
  - University Children's Hospital, Münster
  - Children's Hospital, Rostock
- Semmelweis University, Budapest, Hungary
- Italy (6):
  - S. Orsola-Malphighi Hospital, Bologna
  - Istituto Giannina Gaslini, Genova
  - Fondazione OSP Maggiore Policlinico, Milan
  - University of Padova, Padua
  - Bambino Gesu, Rome
  - Regina Margherita Children's Hospital, Torino
- Vilnius University Children's Hospital, Vilnius, Lithuania
- Poland (4):
  - Medical University Gdansk, Gdansk
  - University Children's Hospital, Krakow
  - Clinic of Pediatrics, Szczecin
  - Children's Memorial Health Institute, Warsaw
- Hospital Sao Joao, Porto, Portugal
- University Children's Hospital, Belgrade, Serbia
- Karolinska University Hospital, Stockholm, Sweden
- Switzerland (2):
  - Inselspital, Bern
  - University Children's Hospital, Zurich
- Turkey (Türkiye) (15):
  - Cukurova Universitesi, Adana
  - Ankara University of Medicine, Ankara
  - Hacettepe Medical Faculty, Ankara
  - Gazi University Hospital, Ankara
  - Baskent University, Faculty of Medicine, Ankara
  - Diskapi Childrens Hospital, Ankara
  - Sami Ulus Childrens Hospital, Ankara
  - Cerrahpasa Tip Fakultesi, Istanbul
  - Istanbul Medical Faculty, Istanbul
  - Bakirkoy Children's Hospital, Istanbul
  - Goztepe Educational and Research Hospital, Istanbul
  - Haseki Educational and Research Hospital, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Sisli Educational and Research Hospital, Istanbul
  - Ege University, Izmir
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- See also: Click here for more information about this study: 4C-Study — http://www.4C-study.org